CLINICAL TRIAL: NCT02339116
Title: FIRST-LINE FOLFOXIRI PLUS BEVACIZUMAB FOLLOWED BY REINTRODUCTION OF FOLFOXIRI PLUS BEVACIZUMAB AT PROGRESSION Versus FOLFOX PLUS BEVACIZUMAB FOLLOWED BY FOLFIRI PLUS BEVACIZUMAB AT PROGRESSION IN FIRST- AND SECOND-LINE TREATMENT OF UNRESECTABLE METASTATIC COLORECTAL CANCER.
Brief Title: Folfoxiri Plus Bev Followed by Reintroduction of Folfoxiri Plus Bev at Progression Versus Folfox Plus Bev Followed by Folfiri Plus Bev in mCRC
Acronym: TRIBE2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIBE2
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Oxaliplatin; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Folfoxiri/bev --> folfoxiri/bev (Experimental): FOLFOXIRI plus bev (to be repeated every 2 weeks for a maximum of 8 cycles):
  Bevacizumab 5 mg/kg iv over 30 minutes, day 1 Irinotecan 165 mg/sqm iv over 60 minutes, day 1 Oxaliplatin 85 mg/sqm iv over 2 hours, day 1 L-Leucovorin 200 mg/sqm iv over 2 hours, day 1 5-fluorouracil 3200 mg/sqm 48 h-continuous infusion, starting on day 1 At the time of disease progression, patients will re-introduce FOLFOXIRI plus bev at the same doses and schedule previously tolerated, for a maximum of 8 cycles. If no progression occurs during FOLFOXIRI plus bev, patients will receive maintenance 5-FU/LV plus bev at the same dose used in the last cycle of the induction treatment.
  Interventions: Drug: fluoruracil; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Bevacizumab
- folfox/bev-->folfiri/bev (Active Comparator): mFOLFOX-6 plus bev (to be repeated every 2 weeks for a maximum of 8 cycles) Bevacizumab 5 mg/kg iv over 30 minutes, day 1 Oxaliplatin 85 mg/sqm iv over 2 hours, day 1 L-Leucovorin 200 mg/sqm iv over 2 hours, day 1 5-fluoruracil 400 mg/sqm iv bolus, day 1 5-fluoruracil 2400 mg/sqm 48 h-continuous infusion, starting on day 1
  At the time of disease progression patients will receive FOLFIRI plus bev (to be repeated every 2 weeks for a maximum of 8 cycles):
  Bevacizumab 5 mg/kg iv over 30 minutes, day 1 Irinotecan 180 mg/sqm iv over 2 hours, day 1 L-Leucovorin 200 mg/sqm iv over 2 hours, day 1 5-fluoruracil 400 mg/sqm iv bolus, day 1 5-fluoruracil 2400 mg/sqm 48 h-continuous infusion.
  Interventions: Drug: fluoruracil; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Bevacizumab

INTERVENTIONS:
Drug: fluoruracil
Drug: Oxaliplatin
Drug: Irinotecan
Drug: Bevacizumab

SUMMARY:
Bev improves the efficacy of first-line chemotherapy in unresectable mCRC. In the phase III TRIBE trial upfront FOLFOXIRI plus bev provided a significant advantage in terms of PFS and RR compared to FOLFIRI plus bev. A trend toward better OS was also evidenced. The second-line treatment was at investigator's choice. A manageable increase in diarrhea, mucositis and neutropenia was reported, while no differences in febrile neutropenia, serious adverse events and toxic deaths were evidenced.

A growing amount of data support the clinical relevance of achieving an early and deep tumor shrinkage.

Phase III TML and BEBYP trials demonstrated that the continuation of bev beyond disease progression combined with a switched chemotherapy regimen provided a significant advantage in terms of OS and PFS.

Based on recent evidences, the partial interruption of the upfront "induction" chemotherapy before disease progression and the prosecution of bev until disease progression as maintenance treatment is a valid strategy in the treatment of mCRC.

On the basis of these considerations, a first-line doublet plus bev followed by a second-line switched doublet (from oxaliplatin to irinotecan and viceversa) plus bev should be considered a standard option for mCRC patients. Only retrospectively collected data are currently available about the efficacy of first-line FOLFOXIRI plus bev followed by second-line rechallenge with FOLFOXIRI plus bev. We therefore designed the present phase III randomized trial of first-line FOLFOXIRI plus bev followed by reintroduction of FOLFOXIRI plus bev at progression versus FOLFOX plus bev followed by FOLFIRI plus bev at progression in first- and second-line treatment of unresectable mCRC patients.

ELIGIBILITY:
Main Inclusion Criteria:

Histologically proven diagnosis of colorectal cancer Initially unresectable metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease At least one measurable lesion according to RECIST1.1 criteria Availability of a tumoral sample Male or female of 18-75 years of age ECOG PS < or = 2 if aged < 71 years, ECOG PS = 0 if aged 71-75 years Life expectancy of at least 12 weeks Previous adjuvant chemotherapy allowed only if with fluoropyrimidine monotherapy and more than 6 months elapsed between the end of adjuvant and first relapse Neutrophils >1.5 x 109/L, Platelets >100 x 109/L, Hgb >9 g/dl Total bilirubin 1.5 time the upper-normal limits (UNL) of the normal values and ASAT (SGOT) and/or ALAT (SGPT) <2.5 x UNL (or <5 x UNL in case of liver metastases) alkaline phosphatase <2.5 x UNL (or <5 x UNL in case of liver metastases) Creatinine clearance >50 mL/min or serum creatinine 1.5 x UNL Urine dipstick of proteinuria <2+. Patients discovered to have 2+ proteinuria on dipstick urinalysis at baseline, should undergo a 24-hour urine collection and must demonstrate <1 g of protein/24 hr Will and ability to comply with the protocol Written informed consent to study procedures and to molecular analyses -

Main Exclusion Criteria:

Radiotherapy to any site within 4 weeks before the study Previous adjuvant oxaliplatin-containing chemotherapy Previous treatment with bevacizumab Untreated brain metastases or spinal cord compression or primary brain tumours History or evidence upon physical examination of CNS disease unless adequately treated Symptomatic peripheral neuropathy > 2 grade NCIC-CTG criteria Serious, non-healing wound, ulcer, or bone fracture Evidence of bleeding diathesis or coagulopathy Uncontrolled hypertension and prior histor of hypertensive crisis or hypertensive encephalopathy Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of study enrolment Any previous venous thromboembolism > NCI CTCAE Grade 3 History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to the first study treatment.

Current or recent (within 10 days prior to study treatment start) ongoing treatment with anticoagulants for therapeutic purposes Chronic, daily treatment with high-dose aspirin (>325 mg/day) Treatment with any investigational drug within 30 days prior to enrollment or 2 investigational agent half-lives (whichever is longer) Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Estimated)
Dates: Start 2015-02-26 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival 2 (PFS2) | from randomization to the first of the following events: a) death; b) disease progression on any treatment given after 1st progression, up to 18 months after last patient last visit
  PFS2 will be defined as beginning with randomization and ending with the first of the following events: a) death; b) disease progression on any treatment given after 1st progression. For patients that will not receive any treatment within 3 months after 1st progression, PFS2 will be equal to PFS. The determination of disease progression will be based on investigator-reported measurements. Disease status will be evaluated according to RECIST 1.1 criteria.
  Censoring rules for PFS2 will be: end of study without PD, loss at follow-up. Curative surgery for metastasis will not result in censoring for PFS2.

SECONDARY OUTCOMES:
Progression free survival (PFS) | from randomization to to the first documentation of objective disease progression or death due to any cause, whichever occurs first, up to 18 months after last patient last visit
  Progression free survival (PFS) is defined as the time from randomization to the first documentation of objective disease progression or death due to any cause, whichever occurs first. PFS will be censored on the date of the last evaluable on study tumor assessment documenting absence of progressive disease for patients who are alive, on study and progression free at the time of the analysis. Alive patients having no tumor assessments after baseline will have time to event censored on the date of randomization
2nd-Progression free survival (2nd-PFS) | from the beginning of the second-line treatment to the documentation of objective disease progression or death due to any cause, whichever occurs first, up to 18 months after last patient last visit
  2nd-Progression free survival (2nd-PFS) is defined as the time from the beginning of the second-line treatment to the documentation of objective disease progression or death due to any cause, whichever occurs first. 2nd-PFS will be censored on the date of the last evaluable on study tumor assessment documenting absence of progressive disease for patients who are alive, on study and 2nd-progression free at the time of the analysis.
Time to failure of strategy (TFS) | from randomization to: death; patient requires a new therapeutic agent; PD on treatment with all agents of the initial strategy; PD during a partial or complete treatment holiday and receives no further therapy within 3 months, up to 18 months after LPLV
  Time to failure of strategy (TFS) is defined as the time time from randomization to the first of the following events: death; patient requires the addition of a new therapeutic agent (i.e. an agent not included in the original strategy); patient experiences disease progression while being treated with all agents that are components of the initial treatment strategy (except for agents which cannot be used because of persistent toxicity or contraindications); or patient experiences disease progression during a partial or complete treatment holiday from initial treatment strategy and receives no further therapy within 3 months. Subjects who did not have an event as stated above while on study will be censored at the last evaluable radiographic assessment date.
Overall survival (OS) | from randomization to the date of death due to any cause up to 18 months after last patient last visit
  Overall survival (OS) is defined as the time from randomization to the date of death due to any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.
Objective Response Rate | Every 8 weeks, up to 18 months after last patient last visit
  percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria, during the induction and the maintenance phases of treatment.
Toxicity Rate | At every cycle of treatment up to the second evidence of PD or up to 18 months after LPLV
  Toxicity Rate is defined as the percentage of patients, relative to the total of enrolled subjects, experiencing a specific adverse event of grade 3/4, according to National Cancer Institute Common Toxicity Criteria (version 4.0), during the induction and the maintenance phases of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Falcone, MD, Study Director — Azienda Ospedaliero Universitaria Pisana, Pisa Italy
Locations (1):
- Polo Oncologico - AOUP, Pisa, PI, Italy

REFERENCES:
- [Derived] Stahler A, Modest DP, Stintzing S, Borelli B, Keller T, Held S, Fischer von Weikersthal L, Muller L, Graeven U, Decker T, Heintges T, Kahl C, Hoppe B, Kiani A, Kaiser F, Schwaner I, Fruehauf S, Karthaus M, Trarbach T, Klauschen F, Horst D, Cremolini C, Heinemann V. Individual Patient Data Meta-Analysis of Consensus Molecular Subtypes as Biomarkers of First-Line Treatment in RAS Wild-Type Metastatic Colorectal Cancer. J Clin Oncol. 2026 Jan;44(1):31-41. doi: 10.1200/JCO-25-00596. Epub 2025 Nov 18. PMID 41252656
- [Derived] Rossini D, Germani MM, Lonardi S, Pietrantonio F, Dell'Aquila E, Borelli B, Allegrini G, Maddalena G, Randon G, Marmorino F, Zaniboni A, Buonadonna A, Boccaccino A, Conca V, Antoniotti C, Passardi A, Masi G, Cremolini C. Treatments after second progression in metastatic colorectal cancer: A pooled analysis of the TRIBE and TRIBE2 studies. Eur J Cancer. 2022 Jul;170:64-72. doi: 10.1016/j.ejca.2022.04.019. Epub 2022 May 17. PMID 35594613
- [Derived] Cremolini C, Antoniotti C, Stein A, Bendell J, Gruenberger T, Rossini D, Masi G, Ongaro E, Hurwitz H, Falcone A, Schmoll HJ, Di Maio M. Individual Patient Data Meta-Analysis of FOLFOXIRI Plus Bevacizumab Versus Doublets Plus Bevacizumab as Initial Therapy of Unresectable Metastatic Colorectal Cancer. J Clin Oncol. 2020 Aug 20:JCO2001225. doi: 10.1200/JCO.20.01225. Online ahead of print. PMID 32816630
- [Derived] Cremolini C, Antoniotti C, Rossini D, Lonardi S, Loupakis F, Pietrantonio F, Bordonaro R, Latiano TP, Tamburini E, Santini D, Passardi A, Marmorino F, Grande R, Aprile G, Zaniboni A, Murgioni S, Granetto C, Buonadonna A, Moretto R, Corallo S, Cordio S, Antonuzzo L, Tomasello G, Masi G, Ronzoni M, Di Donato S, Carlomagno C, Clavarezza M, Ritorto G, Mambrini A, Roselli M, Cupini S, Mammoliti S, Fenocchio E, Corgna E, Zagonel V, Fontanini G, Ugolini C, Boni L, Falcone A; GONO Foundation Investigators. Upfront FOLFOXIRI plus bevacizumab and reintroduction after progression versus mFOLFOX6 plus bevacizumab followed by FOLFIRI plus bevacizumab in the treatment of patients with metastatic colorectal cancer (TRIBE2): a multicentre, open-label, phase 3, randomised, controlled trial. Lancet Oncol. 2020 Apr;21(4):497-507. doi: 10.1016/S1470-2045(19)30862-9. Epub 2020 Mar 9. PMID 32164906
- [Derived] Cremolini C, Marmorino F, Loupakis F, Masi G, Antoniotti C, Salvatore L, Schirripa M, Boni L, Zagonel V, Lonardi S, Aprile G, Tamburini E, Ricci V, Ronzoni M, Pietrantonio F, Valsuani C, Tomasello G, Passardi A, Allegrini G, Di Donato S, Santini D, Falcone A; all the investigators of the Gruppo Oncologico del Nord Ovest. TRIBE-2: a phase III, randomized, open-label, strategy trial in unresectable metastatic colorectal cancer patients by the GONO group. BMC Cancer. 2017 Jun 9;17(1):408. doi: 10.1186/s12885-017-3360-z. PMID 28599628